CLINICAL TRIAL: NCT06345417
Title: Impact of Transfusions and Patient Blood Management on Morbidity and Mortality in Severe Anemia
Brief Title: Outcomes of Patient Blood Management in Severely Anemic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Helios Klinik Gotha/Ohrdruf (Other)
Collaborators: HELIOS Hospital, Erfurt, Germany (Other)
Responsible Party: Principal Investigator, Petra Seeber, Principal Investigator, Helios Klinik Gotha/Ohrdruf
Other Study IDs: O-PBM1
Record Dates: First submitted 2024-02-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Severe Anemia
Keywords: patient blood management; blood transfusion
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PBM only: Participants in study group 1 receive full PBM while they opted not to receive transfusions.
  Full PBM included an individualized, structured approach to detection and management of anemia, bleeding and coagulopathy. PBM is provided in a timely manner.
  Interventions: Other: Patient Blood Management (PBM)
- PBM with transfusion: Participants in the study group 2 receive partial PBM together with transfusions when deemed necessary. Transfusions are given by physicians encouraged to use a restrictive transfusion strategy. PBM is delivered to patients at a convenient time, resorting to a set of standard PBM measures rather than individualized care.
  Interventions: Other: Patient Blood Management (PBM); Biological: Allogeneic transfusion
- Transfusion only: The control group is treated in an environment where PBM is not implemented and transfusion is the standard therapy for severe anemia.
  Interventions: Biological: Allogeneic transfusion

INTERVENTIONS:
Other: Patient Blood Management (PBM) — PBM is a strategy to manage the participant's own blood. Its focus is on anemia, bleeding and coagulation management.
  Groups: PBM only; PBM with transfusion
Biological: Allogeneic transfusion — Anemia is treated by administering donor red cells, and bleeding or coagulopathy by plasma, platelets or other donor blood products.
  Groups: PBM with transfusion; Transfusion only

SUMMARY:
The goal of this observational cohort study is to compare patients with very low red blood counts who receive different therapy. Its main question[s] it aims to answer are:

* Which group of patients dies more frequent: Patients who receive patient blood management only, patients who receive patient blood management and transfusions or patients who receive only transfusions?
* Among these groups: which group of patients has more complications during hospital stay? Patients will either receive patient blood management, which is the management of anemia, bleeding and coagulation problems, will receive transfusions, that is, blood from other people, or a mix of both.

DETAILED DESCRIPTION:
Background:

There seems to be a clear relationship between hemoglobin level and inhospital morbidity and mortality. To mitigate negative effects of lower hemoglobin levels, that is, anemia, transfusions are given when the hemoglobin level of the patient reaches a point deemed detrimental by the treating health care personnel. Patient Blood Management (PBM) adds to the armamentarium of anemia therapy, starting typically well before transfusions are given, and sometimes beyond this point. PBM utilizes medical strategies to enhance the patients own red cell mass and to alleviate the ill effects of disease and bleeding on hematopoesis and homeostasis.

Objective:

The objectives of the present study is to investigate the effects of 2 different management strategies of severe anemia, namely PBM exclusively or PBM with transfusion therapy, and compare them to standard transfusion therapy as regards inhospital mortality and morbidity.

Hypothesis: It is hypothesized that severely anemic participants who received a combination of PBM and restrictive transfusion regime would have a lower mortality and less complications than participants receiving a liberal transfusion therapy without PBM, while participants not being transfused at all will have increased mortality and morbidity.

Setting: The study will be performed at HELIOS Klinikum Gotha (HKG) and Helios Klinikum Erfurt (HKE) which are two neighboring hospitals with overlapping personnel, purchasing, IT departments and standard operating procedures. Both hospitals offer basic, advanced and specialist care to their communities. HKG offers PBM to their patients, while HKE does not.

Data sources: Data will be sourced from the hospital information systems of HKG and HKE.

Diseases are coded with the ICD-10-GM (International Code of Diseases, Version 10, Germany) and procedures using the OPS code (Procedure Key, analogous to the International Code of Procedures).

Participants: All adult patients treated between 1.6.2008 and 31.12.2020 in HKG and HKE will be eligible for enrollment when they were treated by a specialty that both hospitals offer and suffer from severe anemia, defined as a nadir hemoglobin of < 8 g/dL.

Interventions:

Study group 1: Participants in this group received full PBM measures as clinically appropriate, but were not transfused at all.

Study group 2: Participants in this group received convenience measures of PBM and were transfused as deemed necessary in an environment where a restrictive transfusion strategy is encouraged.

Control:

The control group was treated without systematic PBM offered to patients and transfusions were the only standard of care for severely anemic patients.

Outcome:

Primary outcome is inhospital mortality. Secondary outcomes are morbidity measures, such as acute myocardial infarction, blood stream infection, cerebrovascular accident, transfusion complications, readmission rates, etc.

Study design:

This is a dual-center, retrospective observational cohort study. Reporting of results will be performed in line with the REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement extension of the STrengthening the Reporting of OBservational studies in Epidemiology (STROBE) statement.

The study will be guided by a study protocol with an attached statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* adult
* nadir hemoglobin < 8 g/dL

Exclusion Criteria:

* treatment in a non-comparable specialty
* transfer from hospital in the first 6 h after arrival
* requesting PBM / transfusion-free therapy but not offered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all hospitalized participants admitted to Helios Klinikum Gotha and Erfurt between 2008 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of dead participants at the end of hospitalization (inhospital mortality) | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Death at discharge from hospital

SECONDARY OUTCOMES:
Number of participants with surgical wound complications | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Number of participants with a documented presence of surgical wound complications (according to pre-specified ICD list)
Number of participants with a documented acute myocardial infarction | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Acute myocardial infarction (as documented by increase in troponin in conjunction with AMI diagnose)
Number of participants suffering renal injury | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Renal injury (according to RIFLE criteria)
Number of days spent in hospital (Length of stay in hospital) | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Length of stay in hospital, calculated in days
Number of participants readmitted to the studied hospital | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Readmission within 30 days
Number of participants with a documented transfusion reaction | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Transfusion reactions (according to ICD codes T80.3 and T80.4)
Number of participants receiving an allogeneic transfusion | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Transfusion rates per admission, calculated for red blood cells, platelets, plasma
Number of participants treated in an intensive care ward | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Indicator whether or not the participant was treated in an intensive care unit
Number of participants with documented respiratory complications | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Respiratory complications as documented by ventilation support rate (per admission)

CONTACTS AND LOCATIONS:
Overall Officials: Petra Seeber, Principal Investigator — HELIOS Klinikum Gotha
Locations (2):
- Germany (2):
  - Helios Klinikum, Erfurt, Thuringia
  - Helios Klinikum, Gotha, Thuringia

IPD SHARING:
Plan to Share IPD: No